CLINICAL TRIAL: NCT05158491
Title: Safety, Tolerability and Preliminary Efficacy of JK1201I in Patients With Small Cell Lung Cancer
Brief Title: Safety, Tolerability and Preliminary Efficacy of JK1201I in Patients With SCLC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: JenKem Technology Co., Ltd. (Industry)
Collaborators: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: JK-1201I-201
Record Dates: First submitted 2021-11-16; First posted 2021-12-15 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Small Cell Lung Cancer (SCLC)
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — etirinotecan pegol

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 180 mg/mm2 (Active Comparator): Subjects will be dosed at 180 mg/mm2 level.
  Interventions: Drug: JK-1201I
- 220 mg/mm2 (Active Comparator): Subjects will be dosed at 220 mg/mm2 level.
  Interventions: Drug: JK-1201I
- 260 mg/mm2 (Active Comparator): Subjects will be dosed at 260 mg/mm2 level.
  Interventions: Drug: JK-1201I
- 300 mg/mm2 (Active Comparator): Subjects will be dosed at 300 mg/mm2 level.
  Interventions: Drug: JK-1201I

INTERVENTIONS:
Drug: JK-1201I — JK-1201I will be given every 3 weeks, maximum of 4 treatment cycle.
  Other Names: PEG-Irinotecan

SUMMARY:
The purpose of this clinical trial is to evaluate the safety, tolerability and primary efficacy of JK-1201I in patients with small cell lung cancer (SCLC)

DETAILED DESCRIPTION:
This study is a multi-center, open labeled, single, -combined, with multiple dose escalation trial.

The trial consists of dose escalation phase and dose expansion phase; Dose escalation phase: based on the earlier studies, 3 more patients will be added to the 180mg/m2 dose group. The follow-up dose group will adopt the "3+3" design, with 3-6 subjects in each group; include 3 preset dose levels, 220mg/m2, 260mg/m2 and 300mg/m2, respectively. Each subject will receive only one corresponding dose. After the completion of single dose and 21-day DLT observation period, Safety is assessed by the investigator and sponsor, and if the safety evaluation results is favorable, subject will continue to receive the same level of testing compound. Each patient will receive maximum of 4 cycle of treatments.

Dose expansion stage: according to the results of the dose increasing stage, dose groups will be selected for expansion. It is expected that 2 to 3 dose groups will enter the expansion stage, and the total number of participants in each dose group will be 20, and a total of 4 cycles of drug administration will be given to each subject.

ELIGIBILITY:
Inclusion Criteria:

1. Between the age of 18 to 70, male or female;
2. Diagnosed having SCLC via either histology or cytology;
3. Extensive small-cell lung cancer with recurrence or progression within ≤6 months from the end of first-line therapy;
4. At least one measurable lesion (non-intracranial, non-measurable after radiotherapy) according to RECIST version 1.1;.
5. ECOG-PS score is 0-1;
6. Expected survival time ≥12 weeks;
7. Have faverable organ and hematopoietic function, with no serious abnormality of heart, lung, liver or kidney function or immune deficiency according to laboratory tests:
8. Fertile male subjects and female subjects of reproductive age who are willing to take effective non-drug contraceptive measures from signing the informed consent form until 6 months after the last administration of the study drug. Blood pregnancy test results of women of childbearing age must be negative within 7 days before the first trial drug administration.
9. Voluntarily participate in the clinical study and sign the informed consent

Exclusion Criteria:

1. Have a previous history of allergy, or are known to be severely allergic to either JK1201I or its excipients;
2. Previous treatment with topoisomerase I inhibitor (such as irinotecan, topotecan, etc.);
3. At the first use of the drug in this study, other anti-tumor chemotherapy or immunotherapy was stopped for < 4 weeks;
4. CYP3A4 strong inducer was used within 2 weeks before the first administration, or CYP3A4 suppressor or UGT1A1 suppressor was used within 1 week;
5. Patients with clinically serious gastrointestinal dysfunction (positive fecal ocidiocytic blood and severe gastrointestinal bleeding, gastrointestinal infection, obstruction or grade 1 or above diarrhea (increase of stool number ≥4 times per day));
6. Complicated with symptomatic brain metastasis, meningeal metastasis, spinal tumor invasion, spinal cord compression; Superior vena cava syndrome, obstructive atelectasis, and bone metastasis with local symptoms that may require non-medical treatment such as radiotherapy/surgery/endoscopic therapy/interventional therapy;
7. For patients with brain metastasis (the distance from the end of whole brain radiotherapy to the first dose ≤7 days, and the distance from the end of SBRT radiotherapy to the first dose ≤3 days);
8. Patients with severe heart disease within 6 months prior to enrollment, such as unstable angina, heart failure (New York Heart Association Heart function classification > Class II), coronary angioplasty or stenting, deep vein thrombosis, myocardial infarction, etc.; Or other diseases that may affect the subject's safety, such as deep vein thrombosis, stroke, stroke (except caval infarction), poorly controlled active bleeding or known bleeding constitution, etc.);
9. Had a serious pulmonary disease, such as pulmonary fibrosis, active pulmonary tuberculosis, pulmonary hypertension, etc., within 6 months prior to inclusion;
10. Other malignant tumors occurred within 5 years before enrollment, except carcinoma in situ of the cervix, squamous cell carcinoma of the skin or basal cell carcinoma which had been treated for radical treatment before;
11. UGT1A1 suppressor (azanavir, giferozil, etc.) was used or had been used in combination drugs or within 7 days prior to the treatment of the study drugs;
12. large amounts of pleural effusion and ascites needed to be treated (continuous pleural and abdominal effusion > 1000ml within 1 week);
13. Toxicity of previous anti-tumor therapy (including chemotherapy/radiotherapy, surgical therapy, targeted therapy, immunotherapy, Chinese herbal therapy, endocrine therapy or other anti-tumor therapy) has not recovered (grade 1 or above as assessed by CTCAE version 5.0, Except for hair loss, alkaline phosphatase, glutamyltranspeptidase (GGT), or subjects eligible for inclusion after discussion with the investigator and sponsor);
14. Subjects with severe infection within 4 weeks before the first medication, including but not limited to those with infectious complications, bacteremia and severe pneumonia requiring hospitalization;
15. Pregnant or breast-feeding women;
16. Presence of human immunodeficiency virus (HIV) or active hepatitis b (HBsAg positive and HBV-DNA titer ≥1x103 copy number /mL or 200IU/ mL;
17. Subjects who have participated in other clinical trials within 4 weeks prior to obtaining informed consent;
18. Have a clear history of mental disorders;
19. Subjects considered unsuitable for the study by the investigator for other reasons.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2021-11-11 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
To determine dose limited toxicity (DLT) of JK-1201I in patients with SCLC. | 21days
  Dose limited toxicity in SCLC patients will be determined. DLT is defined as: 1..Grade 4 neutropenia (ANC) reduction lasts ≥3 days; or grade 3 ANC reduction with fever (ANC <1000 / mm3 with oral temperature single measurement> 38.3 ℃ or ≥38.0 ℃ for 1 hour)； 2. Grade 3 thrombocytopenia (25×109/L≤ platelet count < 50×109/L) with obvious clinical bleeding symptoms, or grade 4 thrombocytopenia (with or without obvious clinical bleeding symptoms); 3. Other grade 4 hematological toxicity； 4. Grade 3 and above non-hematological toxicity； 5. Hair loss, fatigue, except for those with grade 3 nausea, vomiting, and diarrhea without maximum symptomatic supportive treatment.
To determine the maximum tolerance dose level of JK-1201I in patients with SCLC. | 21days
  MTD is defined as the highest dose that can be given without causing any adverse side effects according to CTCAE v5.0.

SECONDARY OUTCOMES:
To measure the highest plasma concentrations of JK-1201I in patients with SCLC. | 21 days
  The maximum concentration (Cmax) will be measured and compared across different groups.
To determine the exposure levels of JK-1201I in SCLC patients | 21 days
  The area under the plasma concentration versus time curve（AUC）will be compared across different groups.
To examine the primary efficacy of JK-1201I in treating patients with SCLC. | 21days
  Evaluation Criteria In Solid Tumors (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), at least a 30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.

CONTACTS AND LOCATIONS:
Overall Officials: Xuan Zhao, Ph.D., Study Chair — JenKem Technology Co., Ltd.
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No